CLINICAL TRIAL: NCT01052831
Title: Randomized, Double-blind, Placebo-controlled Study of Naltrexone for Impulse Control Disorders in Parkinson's Disease
Brief Title: Naltrexone for Impulse Control Disorders in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Daniel Weintraub, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 810624
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Results first posted 2015-06-22 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-07

CONDITIONS: Impulse Control Disorder; Parkinson Disease
Keywords: Compulsive Gambling; Compulsive Buying; Compulsive Shopping; Compulsive Eating; Hypersexuality; Dopamine Agonists; Mirapex; Pramipexole; Requip; Ropinirole; Impulse Control Disorders
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders; Parkinson Disease; Gambling; Food Addiction; Compulsive Sexual Behavior Disorder | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naltrexone (Active Comparator): For the first four weeks of the study, participants were administered naltrexone at 50mg per day. Participants not in response at week 4 were increased to 100mg per day for the remaining four weeks of the study.
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): Participants received the placebo treatment which looked identical to active study medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — 50-100 mg qd for 8 weeks
  Other Names: Revia, Vivitrol
  Arms: Naltrexone
Drug: Placebo — 50-100 mg qd for 8 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of naltrexone in reducing ICD symptoms in Parkinson's disease patients taking a dopamine agonist.

DETAILED DESCRIPTION:
Impulse control disorders (ICDs), including compulsive gambling, sexual behavior, buying, and eating, are increasingly recognized as a significant clinical problem in Parkinson's disease (PD), occurring in up to 15% of patients. Dopamine agonist (DA) treatment is thought to be the primary risk factor for the development of ICDs in PD. ICDs often lead to significant impairments in psychosocial functioning, interpersonal relationships, and quality of life. The management of ICDs in the context of PD can be complex. Patients may be reluctant to discontinue DA treatment due to the motor benefits derived from treatment, so patients often have chronic symptoms. Thus, additional treatment approaches are needed.

A medication shown to be efficacious for the treatment of ICDs with minimal impact on parkinsonism would allow many ICD patients to continue on full-dose DA treatment. Naltrexone, a long-acting opioid receptor antagonist, helps in the treatment of alcohol and opioid dependence. In addition, placebo-controlled studies have demonstrated that it helps in the treatment of pathological gambling in the general population. Opioids regulate dopamine pathways in areas of the brain linked with impulse control disorders, and opioid antagonists block opioid receptors in these regions. In this study, 48 PD patients with an ICD will be treated either with naltrexone (50-100 mg/day) or placebo for a period of 8 weeks. The study will assess if naltrexone improves ICD symptoms in PD and is well tolerated. To our knowledge, the proposed study is the first controlled trial of an agent to treat ICDs in PD.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of possible or probable idiopathic Parkinson's disease (PD).
2. Ages 18-85 years.
3. Diagnosis of compulsive gambling, buying, sex behavior, or eating of >2 months duration.
4. Impulse control disorder (ICD) behaviors that began after PD onset and in context of dopamine agonist (DA) treatment.
5. Current stable DA use. Participants must be on a DA for 6 months and on a stable dose (no changes) for 1 month prior to enrolling the in the study.
6. Subjects are capable of giving informed consent, supported by not having significant cognitive impairment based on Montreal Cognitive Assessment score ≥24.
7. Willingness to maintain existing PD pharmacotherapy regimen for the duration of the study.

Exclusion Criteria

1. Active suicide ideation.
2. Anticipated need to initiate antidepressant therapy during the course of the study (must be on a dose in the therapeutic range for at least 2 months. If patient does end up needing to start antidepressant or change antidepressant dose during the course of the study, he/she will be allowed to continue study participation).
3. ICD behaviors so severe that modification of DA treatment is clinically warranted, as judged by PI.
4. Deep brain stimulation surgery in the past year.
5. Evidence for significant liver disease by chart review or patient history (e.g., cirrhosis, chronic hepatitis, liver transplant, or liver cancer).
6. Meeting diagnostic criteria for alcohol or opiate dependence.
7. Meeting diagnostic criteria for Dopamine Dysregulation Syndrome.
8. Use of opioids for pain management.
9. Females that are pregnant, planning to become pregnant, or are breastfeeding will not be included in the study. Females of child bearing potential will need to verify that they are not pregnant by a negative urine pregnancy test.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Weintraub, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Papay K, Xie SX, Stern M, Hurtig H, Siderowf A, Duda JE, Minger J, Weintraub D. Naltrexone for impulse control disorders in Parkinson disease: a placebo-controlled study. Neurology. 2014 Aug 26;83(9):826-33. doi: 10.1212/WNL.0000000000000729. Epub 2014 Jul 18. PMID 25037206

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 26 | 24
Completed | 22 | 23
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Naltrexone: Participants will receive Naltrexone
  Naltrexone: 50-100 mg qd for 8 weeks
- Placebo: Participants will receive placebo treatment
  Placebo: 50-100 mg qd for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.0) | 61.0 (8.2) | 61.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 16 | 6 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 26 | 23 | 49
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Assessed as Very Much Improved or Much Improved Based on the Clinical Global Impression-Improvement (CGI-I) Scale
Description: The Clinical Global Impression-Improvement scale rates total improvement on a 7 point scale:
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse
  A participant scoring a 1 or 2 is considered a responder on the CGI scale. For the change in response status over time, a generalized estimating equation (GEE) model was used.
Time Frame: The CGI-I was administered at Visit 2 (week 2, two weeks after baseline) and Visit 5 (week 8, termination visit 8 weeks after baseline).
Measure: Number; unit: percentage of responders
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 26 | 24
percentage of responders | 54.4 | 33.1

2. Secondary Outcome: Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease - Rating Scale (QUIP-RS)
Description: The Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS) was developed for use in clinical trials and added as a secondary outcome measure for assessment of change in severity of ICD symptoms, to be completed at baseline and end of study only. For the QUIP-RS, scores for each compulsive behavior range from 0 to 16, with a higher score indicating greater severity (frequency) of symptoms. Given that ICD symptoms are frequently comorbid in patients with PD, total QUIP-RS ICD scores (range from 0 to 64) were used to compare overall severity of ICD symptoms. Please note that this measure is reporting a change from baseline.
Time Frame: The QUIP-RS was administered at baseline and the termination visits (Visit 5, 8 weeks after baseline).
Population: A linear mixed-effects model was used to estimate changes in QUIP-RS ICD scores from baseline to termination (visit 5, 8 weeks after baseline). Positive estimated change values represent a decrease in severity (frequency) of symptoms.
Measure: Number (95% Confidence Interval); unit: Change in points on a scale (QUIP-RS)
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 26 | 24
Change in points on a scale (QUIP-RS) | 14.92 [9.89 to 19.96] | 7.55 [2.45 to 12.66]

ADVERSE EVENTS:
Description: A total of 48 patients provided adverse event data.
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 18/24 | 14/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone (N=24) | Placebo (N=24)
Nausea (Gastrointestinal disorders) | 7 (7) | 0 (0)
Dizziness (General disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 5 (5) | 4 (4)
Blood Pressure Change (General disorders) | 6 (6) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No